CLINICAL TRIAL: NCT02879396
Title: Preventing Avoidable Admissions Among Assisted Living Elders (PA4LE)
Brief Title: Preventing Avoidable Admissions Among Assisted Living Elders
Acronym: PA4LE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Jeannie K Lee, Associate Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1608799126
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Aging; Emergencies
Keywords: Older adults; Avoidable admissions; Assisted living home; Emergency service calls; Heading Assisted Living Facilities
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Participants (Experimental): A maximum of 50 participants will be enrolled in the study per the inclusion and exclusion criteria. The participants will be residents of SLH who are 55 years old or older. They will have had one or more EMS calls made, ED visit or hospital admission in the past year, as determined by the incidence report at SLH. The study participants will receive PA4LE program.
  Interventions: Behavioral: PA4LE Program

INTERVENTIONS:
Behavioral: PA4LE Program — 1. Medication self-management including medication reconciliation, therapy recommendations, and education by pharmacist (chronic conditions and medications including Beers Criteria)
  2. Use of a patient-centered health record that helps guide patients through the care process (portable, health and medication record for elders)
  3. Primary care provider and specialist follow-up (patient awareness of discharge action plan and follow-up)
  4. Patient understanding of "red flag" indicators of worsening condition and appropriate next steps
  5. Behavioral interventions - Adherence, Lifestyle modifications, Mindfulness & Lovingkindness meditations to combat anxiety, insomnia and other behavioral symptoms

SUMMARY:
Saint Luke Home (SLH) is a home for low-income seniors who are ≥ 55 years and in need of basic living help in Tucson, Arizona. Reports shows that emergency calls are made from SLH (64 residents) around 60 times each year with emergency department (ED) visits and hospital admissions that follow. In 2014, a total of 70 calls were made, and in 2015, 49 calls. The Director, who is a nurse by training, and staff report that many of these calls are related to medications and may be avoidable. Therefore, we believe we can make a difference and decrease emergency calls, ED visits and hospitalizations that can be avoided with a program to teach the elders and staff at SLH. The program is called Preventing Avoidable Admissions Among Assisted Living Elders (PA4LE) and will consist of a 2-hour session every two weeks including home or clinic visits (elder preference), educational sessions, and staff training.

DETAILED DESCRIPTION:
Saint Luke Home (SLH) is the only nondenominational, nonprofit academic assisted living center (ALC) for low-income seniors who are ≥ 55 years old and in need of supervisory level assistance in Tucson, Arizona. SLH residents have high behavioral health overlay with presence of cognitive decline for some elders. Arizona Center on Aging and University of Arizona Health Sciences have established an academic partnership with SLH. Currently, interprofessional student teams conduct monthly screening clinics at SLH, but these visits are limited to education, simple screening measures, and making general recommendations to the elder's primary care provider via fax. Elders living at SLH have multiple providers for their chronic conditions, and those providers may not be trained in geriatric care.

The documentation from incident reports shows that emergency medical service (EMS) calls are made from SLH (capacity 64) approximately 60 times each year with emergency department (ED) visits and hospital admissions following the incidences. In 2014, a total of 70 calls were made, whereas 49 calls were made in 2015. The Director, who is a nurse by training, and staff reported that many of these calls are medication-related and may be avoidable. As a quality improvement process, a root-cause analysis was conducted by the PharmD fellows interested in geriatric care and research with results reported. From the period of March 2015 to March 2016, a total of 65 calls were made to 911 from SLH that resulted in 39 ED visits and 6 hospitalizations by SLH elders. This was approximately 2 incidences/elder.

We believe forming an interprofessional team to bridge care and decrease EMS calls, ED visits and hospitalizations can make a difference, a program entitled Preventing Avoidable Admissions Among Assisted Living Elders (PA4LE). The interprofessional team will consist of PI (PharmD with board certification in Geriatric Pharmacy), two doctor of pharmacy fellows, Psychiatric nurse practitioner (NP), SLH director (nurse by training), and SLH resident manager. All clinical activities will be supervised by a faculty team of geriatric attendings - Dr. Fain (MD), Dr. Mohler (NP), and Dr. Lee (PI, PharmD). The PA4LE program will consist of bi-weekly, 2-hour sessions, which will include home or clinic visits (elder preference), educational sessions, and staff training at the SLH.

The purpose of the PA4LE program is to prevent EMS calls, ED visits and hospital admissions from avoidable causes and decrease the use of high-risk medications among elders at the SLH. We are modeling the current study intervention in part after the Coleman Care Transitions Model, which is a patient and family-centered care transitions program from hospital to community. The components of the model will be translated into use for ED/Hospital to ALC transitions to avoid EMS calls, ED visits and hospital admissions/readmissions. To identify avoidable causes for admissions, we used the study by Ouslander et al. that determined frequency, causes and costs of potentially avoidable hospitalizations among nursing home residents. A maximum of 50 participants will be enrolled in the study per the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* One or more EMS calls made, ED visit or hospital admission in the past year, as determined by the incidence report at SLH

Exclusion Criteria:

* A score of ≤ 22 out of 30 on the Montreal Cognitive Assessment (MoCA) during initial assessment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
EMS calls | 12 months
  Reduce the number of EMS calls from avoidable causes by high-utilizers (≥ 4 calls) by 50%

SECONDARY OUTCOMES:
ED visits | 12 months
  Reduce the number of ED visits and hospital admissions for avoidable causes by high utilizers (≥ 2/year) by 50%
Beers criteria medications | 12 months
  Reduce the number of Beers Criteria medications (inappropriate for older adults) by 15% among high-users (≥2)

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie K Lee, PharmD, Principal Investigator — University of Arizona
Locations (1):
- St. Luke's Home, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No